CLINICAL TRIAL: NCT02690961
Title: Randomized, Double-blind Placebo-controlled Phase I Study to Assess Safety, Tolerance，Pharmacokinetics of Multiple-dose Kukoamine B Mesilate in Healthy Volunteers
Brief Title: Study of Multiple-dose Kukoamine B Mesilate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Chasesun Pharmaceutical Co., LTD (Industry)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-KB103; ChiCTR-TRC-14005111 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2016-02-05; First posted 2016-02-24 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Kukoamine B Mesilate 0.06mg/kg (Experimental): Dose Escalation: Kukoamine B Mesilate 0.06mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.12mg/kg (Experimental): Dose Escalation: Kukoamine B Mesilate 0.12mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Kukoamine B Mesilate 0.24mg/kg (Experimental): Dose Escalation: Kukoamine B Mesilate 0.24mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: Kukoamine B Mesilate
- Placebo 0.06mg/kg (Experimental): Dose Escalation: placebo 0.06mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: placebo multiple doses
- Placebo 0.12mg/kg (Experimental): Dose Escalation: placebo 0.12mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: placebo multiple doses
- Placebo 0.24mg/kg (Experimental): Dose Escalation: placebo 0.24mg/kg multiple-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Interventions: Drug: placebo multiple doses

INTERVENTIONS:
Drug: Kukoamine B Mesilate — Kukoamine B Mesilate or placebo single-dose and intravenous(IV) drip for 1 hour in healthy volunteers.
  Arms: Kukoamine B Mesilate 0.06mg/kg; Kukoamine B Mesilate 0.12mg/kg; Kukoamine B Mesilate 0.24mg/kg
Drug: placebo multiple doses
  Arms: Placebo 0.06mg/kg; Placebo 0.12mg/kg; Placebo 0.24mg/kg

SUMMARY:
The purpose of this study is to assess safety, tolerance and pharmacokinetics of Multiple-dose Kukoamine B Mesilate in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male or female, each sex ratio does not exceed 2/3;
2. 18-45 years (including upper and lower limit), the general situation is good;
3. Body mass index (BMI) in 19-28 (including upper and lower limit of the range), bodyweight（BW）≥ 50kg (female) and 60kg (male);
4. Nearly half of the year, no child care program and agreed to take effective measures to contraception during the study period, women of childbearing age blood pregnancy test was negative;
5. Subjects to fully understand the purpose, properties, method and reactions may occur of test drug trials.Voluntarily signed the informed consents, and agreed to abide by the requirements of clinical protocols.

Exclusion Criteria:

1. Primary disease in important organs;
2. Mental or physical disability;
3. Familial hereditary disease;
4. Screening supine blood pressure (after 5 minutes of rest) systolic or diastolic blood pressure greater than 90-140 millimeters of mercury(mmHg), beyond the scope of 50-90 millimeters of mercury(mmHg), Or pulse (HR) beyond 50bpm-100bpm;
5. Abnormal results of any clinically meaningful physical examination, vital signs, ECG or clinical laboratory;
6. History of immunodeficiency diseases, including HIV antibody positive;
7. Detection of antibody positive, hepatitis B surface antigen or antibody to hepatitis C / syphilis positive;
8. Alcohol and drug abusers;
9. Who is addicted to alcohol and tobacco (drinking 14 units of alcohol per week: 1 unit = beer 285 ml, or liquor 25 ml, or wine 1 cup. numbers of daily smoking ≥ 5) and / or not smoking and drinking in the test period;
10. Any discharge period may affect the study drug, or in the past 3 months participated in any drug clinical trials;
11. Before entering the group 4 weeks using any prescription drugs before entering the group, or use of any non prescription drugs within 2 weeks (vitamins, herbal tonics, etc.), or into the group within 2 weeks before taking effect of drug metabolizing enzymes in food, such as grapefruit or grapefruit drink. Can the use of acetaminophen, but must record report in case report form（CRF）;
12. The last 3 months had a history of blood donation or significant blood loss (more than 400ml);
13. There are drugs, the clinical significance of the history of food allergy and atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known drug to test drugs or similar drug allergy test;
14. Lactating women, pregnant women or unable to take effective contraceptive measures;
15. Researchers believe that participants not suitable to take the test for other factors .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events. | 14 days
  adverse event, physical examination, monitoring of vital signs, Laboratory examination, electrocardiogram(ECG).

SECONDARY OUTCOMES:
Pharmacokinetic parameters(Maximum Plasma Concentration [Cmax]) | the first day,the sixth day(before the three injections from bottom),the seventh day
  before the first injecting(omin); after starting the first injecting 30min;ending the first injecting instantly,1h,3h,6h,8h,12h,16h,23h;before the three injections from bottom,after starting the last injecting 30min,ending the last injecting instantly,1h,3h,6h,8h,12h,16h,23h.

OTHER OUTCOMES:
Pharmacokinetic parameters(Area Under Curve [AUC]) | the first day,the sixth day(before the three injections from bottom),the seventh day
  before the first injecting(omin); after starting the first injecting 30min;ending the first injecting instantly,1h,3h,6h,8h,12h,16h,23h;before the three injections from bottom,after starting the last injecting 30min,ending the last injecting instantly,1h,3h,6h,8h,12h,16h,23h.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Chen, Study Director — Tianjin Chasesun Pharmaceutical Co., LTD
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao Q, Liu H, Wang Z, Wang T, Cui C, Wang H, Li L, Zhong W, Jiang J, Dong K, Chen S, Jin C, Hu P. Safety, Tolerability, and Pharmacokinetics of Kukoamine B in Healthy Volunteers: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Phase I Study. Adv Ther. 2023 Jul;40(7):3186-3198. doi: 10.1007/s12325-023-02521-1. Epub 2023 May 26. PMID 37233875